CLINICAL TRIAL: NCT06018935
Title: A Cohort Establishment Study of Total Management of Ovarian Cancer (Including Fallopian Tube Cancer and Primary Peritoneal Cancer)
Brief Title: A Cohort Establishment Study of Total Management of Ovarian Cancer
Status: Recruiting | Type: Observational
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Dengfeng Wang, Deputy chief, Sichuan Cancer Hospital and Research Institute
Other Study IDs: LCATM202304
Record Dates: First submitted 2023-08-10; First posted 2023-08-31 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Tumor of Female Reproductive System; Ovarian Cancer
Keywords: Ovarian cancer; Cohort study; Whole-process management
MeSH Terms: conditions — Genital Neoplasms, Female; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
A cohort establishment study of total management of ovarian cancer (including fallopian tube cancer and primary peritoneal cancer).

DETAILED DESCRIPTION:
1. To investigate the effects of surgery, chemotherapy, maintenance therapy and related factors on the prognosis and quality of life of patients with ovarian cancer (including fallopian tube cancer and primary peritoneal cancer);
2. To study the postoperative recovery of patients with ovarian cancer (including fallopian tube cancer and primary peritoneal cancer), perioperative complications, adverse reactions after chemotherapy, adverse reactions during targeted drug maintenance therapy, and explore possible effective preventive measures;
3. The prognostic factors of ovarian cancer (including fallopian tube cancer and primary peritoneal cancer) were analyzed;
4. To study the efficacy and safety of PARPi in clinical application in patients with ovarian cancer (including fallopian tube cancer and primary peritoneal cancer).

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with ovarian cancer (including fallopian tube cancer, primary peritoneal cancer) and intended to be treated in our hospital;
2. Can cooperate with later follow-up.

Exclusion Criteria:

1. Patients with other malignant tumors or previous history of other malignant tumors;
2. Have cognitive impairment.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with ovarian cancer (including fallopian tube cancer, primary peritoneal cancer) and intended to be treated in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Progress Freesurvival (PFS) | Average six months after study completion.
  The time from the start of treatment until the patient progresses further or dies.
Overall Survival (OS) | Average six months after study completion.
  Measure the time from the start of treatment to the time of death.

SECONDARY OUTCOMES:
Occurrence of adverse reactions | Average six months after study completion.
  All adverse events were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital, Chengdu, China

IPD SHARING:
Plan to Share IPD: No